CLINICAL TRIAL: NCT02677584
Title: Prophylactic Versus Therapeutic Caffeine for Apnea of Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Nehad Nasef, Principle Invistigator, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R / 15.06.75
Record Dates: First submitted 2016-01-03; First posted 2016-02-09 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Apnea
Keywords: caffeine; apnea; preterm infant
MeSH Terms: conditions — Apnea; Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic caffeine citrate (Active Comparator): Prophylactic caffeine (group1) will be defined as caffeine prescribed for preterm infant within the first 72 hours of life prior to manifest apnea . patients will be randomly assigned to receive caffeine in loading dose 20 mg/kg (equivalent for 10 mg/kg caffeine base) and maintenance dose 10 mg/kg/day (equivalent for 5 mg/kg caffeine base) .
  Interventions: Drug: Prophylactic caffeine citrate
- Therapeutic caffeine citrate (Active Comparator): Therapeutic caffeine ( group 2 ) will be defined as caffeine prescribed for manifest apnea within or after the first 72 hours of life . patients will be randomly assigned to receive caffeine in loading dose 20 mg/kg (equivalent for 10 mg/kg caffeine base) and maintenance dose 10 mg/kg/day (equivalent for 5 mg/kg caffeine base).
  Interventions: Drug: Therapeutic caffeine citrate

INTERVENTIONS:
Drug: Prophylactic caffeine citrate — Prophylactic caffeine (group1) will be defined as caffeine prescribed for preterm infant within the first 72 hours of life prior to manifest apnea . patients will be randomly assigned to receive caffeine in loading dose 20 mg/kg (equivalent for 10 mg/kg caffeine base) and maintenance dose 10 mg/kg/day (equivalent for 5 mg/kg caffeine base) .
  Arms: Prophylactic caffeine citrate
Drug: Therapeutic caffeine citrate — Therapeutic caffeine ( group 2 ) will be defined as caffeine prescribed for manifest apnea within or after the first 72 hours of life . patients will be randomly assigned to receive caffeine in loading dose 20 mg/kg (equivalent for 10 mg/kg caffeine base) and maintenance dose 10 mg/kg/day (equivalent for 5 mg/kg caffeine base).
  Arms: Therapeutic caffeine citrate

SUMMARY:
Investigators hypothesized that the timing of caffeine administration in either prophylaxis or treatment of apnea of prematurity will affect the apnea response to caffeine

DETAILED DESCRIPTION:
It will be a randomized control trial, patients will be randomly assigned to receive caffeine in a loading dose of 20 mg/kg (equivalent to 10 mg/kg caffeine base) and a maintenance dose of 10 mg/kg/day (equivalent to 5 mg/kg caffeine base) either as a prophylaxis group (1) or therapeutic group (2). Prophylactic caffeine (group 1) will be defined as caffeine prescribed for preterm infants within the first 72 hours of life prior to manifest apnea , therapeutic caffeine ( group 2 ) will be defined as caffeine prescribed for manifest apnea within or after the first 72 hours of life .

Preparation and administration of caffeine will be performed by a Neonatal intensive care unit (NICU) nurse.

Statistical Evaluation:

Statistical analyses will be performed with the Statistical Package for Social Sciences-SPSS version 16 software (SPSS Inc, Chicago, Illinois). For categorical variables, the X2 test will be used. For group comparisons, the Student T test will be used in normal distribution and the Mann-Whitney U test will be used in case of abnormal distribution.

For repeating measurements, variance analyses and Friedman variance analyses will be used. For descriptive statistics, percent, minimum-maximum-median, mean, and standard deviation will be used in accordance with the type and distribution of the variable. A P value <.05 was considered statistically significant. Informed consent will be obtained from parents, and the study will be approved by the local ethical committee.

ELIGIBILITY:
Inclusion Criteria:

* Infants eligible for this study will be newborn infants ≤ 32 weeks with or without a diagnosis of apnea .

Exclusion Criteria:

* Newborn infants with gestational age > 32 weeks.
* Newborn infants with congenital malformations and chromosomal anomalies.
* Newborn infants with apnea of other causes .

Ages: 1 Hour to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2015-03; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Duration of Respiratory Support | 60 days from NICU admission

SECONDARY OUTCOMES:
Days of apnea free | 60 days from NICU admission
length of hospital stay | 60 days from NICU admission
Head ultrasound results | 14 days from NICU admission
  Any grade of intraventricular hemorrhage (IVH); periventricular leukomalacia (PVL)
Necrotizing Enterocolitis | 30 days from NICU admission
  Any stage, according to modified Bell classification
Retinopathy of prematurity | 60 days from NICU admission
  Any stage, according to International classification of retinopathy of prematurity (ICROP)

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, El Dakahlya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dobson NR, Patel RM, Smith PB, Kuehn DR, Clark J, Vyas-Read S, Herring A, Laughon MM, Carlton D, Hunt CE. Trends in caffeine use and association between clinical outcomes and timing of therapy in very low birth weight infants. J Pediatr. 2014 May;164(5):992-998.e3. doi: 10.1016/j.jpeds.2013.12.025. Epub 2014 Jan 23. PMID 24461786
- [Background] Katheria AC, Sauberan JB, Akotia D, Rich W, Durham J, Finer NN. A Pilot Randomized Controlled Trial of Early versus Routine Caffeine in Extremely Premature Infants. Am J Perinatol. 2015 Jul;32(9):879-86. doi: 10.1055/s-0034-1543981. Epub 2015 Jan 21. PMID 25607226